CLINICAL TRIAL: NCT03012932
Title: HPV Self-Sampling for Cervical Cancer Screening Among Lesbian, Bisexual, and Queer (LBQ) Women: A Pilot Study
Brief Title: HPV Self-Sampling for Cervical Cancer Screening Among Lesbian, Bisexual, and Queer (LBQ) Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Julia Seay, Research Assistant Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20161052
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Cervical Cancer Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV Self-sampling (Other): All participants will receive HPV self-sampling intervention. HPV self-sampling is a cervical cancer screening that can be done in private, using a device that is similar to a tampon. This intervention tests for high-risk HPV, the primary cause of cervical cancer. Each participant will complete the intervention one time only.
  Interventions: Behavioral: HPV self-sampling

INTERVENTIONS:
Behavioral: HPV self-sampling — All participants will receive HPV self-sampling intervention. HPV self-sampling is a cervical cancer screening that can be done in private, using a device that is similar to a tampon. This intervention tests for high-risk HPV, the primary cause of cervical cancer. Each participant will complete the intervention one time only.

SUMMARY:
The proposed study will examine the implementation of a Human Papilloma Virus (HPV) self-sampling intervention for under screened LBQ women living in South Florida. The study will enroll participants to receive the self-sampling intervention in community venues. The purpose of this study is to pilot the self-sampler for feasibility and acceptability within this underserved population.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as lesbian, bisexual, or queer woman
* Assigned female sex at birth
* English speaking
* ages 25-65 years
* report not having had a pap smear in the last three years (per USPSTF guidelines)
* if age 30 or over, report not having a pap smear/HPV co-test within the past 5 years (per USPSTF guidelines)

Exclusion Criteria:

* report having had a hysterectomy
* report having history of cervical cancer
* unable to consent
* Pregnant women
* Prisoners

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2018-03-24 (Actual); Study Completion 2018-03-24 (Actual)

PRIMARY OUTCOMES:
HPV Self-sampling uptake | through study completion, up to 1 year
  Percentage of eligible women who complete HPV self-sampling

CONTACTS AND LOCATIONS:
Overall Officials: Julia Seay, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No